CLINICAL TRIAL: NCT00005294
Title: Developmental Sequelae of Severe Chronic Lung Disorders
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 2017; R01HL038193 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-04

CONDITIONS: Bronchopulmonary Dysplasia; Lung Diseases
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Lung Diseases

SUMMARY:
To determine the impact of bronchopulmonary dysplasia (BPD) on childhood development, family functioning, and parental stress.

DETAILED DESCRIPTION:
BACKGROUND:

Bronchopulmonary dysplasia in infancy has been shown to be related to less optimal physical and psychological functioning later in life. Although infants with the disorder increased from 1978 to 1988, little was known about potential developmental problems early in life which might lead to the documented negative sequelae shown in previous research.

DESIGN NARRATIVE:

In this longitudinal study, infants were followed from birth and given standardized assessments of developmental and physical functioning. Demographic, birth, and medical data were collected at baseline through chart review. Standardized questionnaires measuring parental stress and family support were administered to the parents. Infants were followed at eight months, and one, two, and three years at which time parental measures were repeated and standardized assessments made of the children's physical growth, medical status, cognitive, language and behavioral development. Feeding behaviors were assessed through standardized observation and interview at each visit. Data were evaluated descriptively as well as through a series of multivariate analyses of variance with repeated measures.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1989-07; Study Completion 1995-06 (Actual)

REFERENCES:
- [Background] Singer L, Yamashita T, Lilien L, Collin M, Baley J. A longitudinal study of developmental outcome of infants with bronchopulmonary dysplasia and very low birth weight. Pediatrics. 1997 Dec;100(6):987-93. doi: 10.1542/peds.100.6.987. PMID 9374570
- [Background] Singer L, Martin RJ, Hawkins SW, Benson-Szekely LJ, Yamashita TS, Carlo WA. Oxygen desaturation complicates feeding in infants with bronchopulmonary dysplasia after discharge. Pediatrics. 1992 Sep;90(3):380-4. PMID 1518692
- [Background] Singer L, Farkas K, Kliegman R. Childhood medical and behavioral consequences of maternal cocaine use. J Pediatr Psychol. 1992 Aug;17(4):389-406. doi: 10.1093/jpepsy/17.4.389. PMID 1382125
- [Background] Singer LT, Ambuel B, Wade S, Jaffe AC. Cognitive-behavioral treatment of health-impairing food phobias in children. J Am Acad Child Adolesc Psychiatry. 1992 Sep;31(5):847-52. doi: 10.1097/00004583-199209000-00011. PMID 1400116
- [Background] Singer LT, Hill BP, Orlowski JP, Doershuk CF. Medical and social factors as predictors of outcome in infant tracheostomy. Pediatr Pulmonol. 1991;11(3):243-8. doi: 10.1002/ppul.1950110310. PMID 1722034
- [Background] Singer LT, Garber R, Kliegman R. Neurobehavioral sequelae of fetal cocaine exposure. J Pediatr. 1991 Oct;119(4):667-72. doi: 10.1016/s0022-3476(05)82426-6. PMID 1919905
- [Background] Singer LT, Nofer JA, Benson-Szekely LJ, Brooks LJ. Behavioral assessment and management of food refusal in children with cystic fibrosis. J Dev Behav Pediatr. 1991 Apr;12(2):115-20. PMID 2045484
- [Background] Singer LT, Yamashita TS, Hawkins S, Cairns D, Baley J, Kliegman R. Increased incidence of intraventricular hemorrhage and developmental delay in cocaine-exposed, very low birth weight infants. J Pediatr. 1994 May;124(5 Pt 1):765-71. doi: 10.1016/s0022-3476(05)81372-1. PMID 7513757
- [Background] Singer L, Arendt R, Minnes S. Neurodevelopmental effects of cocaine. Clin Perinatol. 1993 Mar;20(1):245-62. PMID 8458168
- [Background] Singer L, Arendt R, Song LY, Warshawsky E, Kliegman R. Direct and indirect interactions of cocaine with childbirth outcomes. Arch Pediatr Adolesc Med. 1994 Sep;148(9):959-64. doi: 10.1001/archpedi.1994.02170090073014. PMID 8075743
- [Background] Singer LT, Davillier M, Preuss L, Szekely L, Hawkins S, Yamashita T, Baley J. Feeding interactions in infants with very low birth weight and bronchopulmonary dysplasia. J Dev Behav Pediatr. 1996 Apr;17(2):69-76. PMID 8727839